CLINICAL TRIAL: NCT02370628
Title: Vertebroplasty In The Treatment Of Acute Fracture Trial (The VITTA Trial)
Brief Title: Vertebroplasty In The Treatment Of Acute Fracture Trial - The VITTA Trial
Acronym: VITTA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: too few participants enrolled and few interested patients in three years
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE14.334
Record Dates: First submitted 2015-02-09; First posted 2015-02-25 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Vertebral Compression Fractures
Keywords: percutaneous vertebroplasty; facet block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous vertebroplasty (PV) (Experimental): The procedure involves percutaneous application of bone cement (polymethylmethacrylate) into collapsed vertebrae.
  Interventions: Procedure: Percutaneous vertebroplasty; Procedure: Facet block
- Facet block (Active Comparator): injection of anti-inflammatory and analgesic drugs
  Interventions: Procedure: Facet block

INTERVENTIONS:
Procedure: Percutaneous vertebroplasty — The procedure involves percutaneous application of bone cement (polymethylmethacrylate) into collapsed vertebrae, and has been used for treatment of patients with osteoporosis who have severe or prolonged pain following vertebral compression fracture, as well as those with painful, aggressive hemangiomas and osteolytic neoplasms.
  In our trial, vertebroplasty shall be performed in two steps:
  * Step 1: facet block
  * Step 2: cement infusion
  Therefore, patients in both arms will undergo Step 1 since our control intervention serves as a routine first part of our active intervention.
  Arms: Percutaneous vertebroplasty (PV)
Procedure: Facet block — A long-acting local anesthetic agent and corticosteroids are injected in the spinal articular facets at the affected level.
  All patients will undergo facet block since it serves as a routine first part to percutaneous vertebroplasty.

SUMMARY:
The VITTA trial is a randomized, controlled, single-blinded, cross-over trial comparing percutaneous vertebroplasty with facet block in patients with acute (<1month) and painful vertebral compression fractures.

The treatment offered for vertebral compression fractures (VCFs) in the interventional arm of the trial is vertebroplasty, which will be performed in accordance with the standardized protocol of the Canadian Association of Radiologists. Patients in the control arm will receive facet block, where a long-acting local anesthetic agent and corticosteroids are injected in the spinal articular facets at the affected level.

DETAILED DESCRIPTION:
Vertebroplasty is a procedure used to stabilize broken vertebrae, the bones that form the spine. This study will evaluate the effectiveness of vertebroplasty for the treatment of acute vertebral fractures.

The VITTA trial is a randomized, controlled, single-blinded, cross-over trial comparing percutaneous vertebroplasty with facet block in patients with acute (<1 month) and painful vertebral compression fractures.

Vertebral compression fractures (VCFs) frequently result in debilitating pain, impaired functional status and bad quality of life. Percutaneous vertebroplasty (PV) is a treatment for VCFs originally developed in France in the late 1980s and first performed in America in the mid-1990s. The procedure involves percutaneous application of bone cement (polymethylmethacrylate) into collapsed vertebrae.

VCFs are a significant public health problem with approximately 750,000 new fractures occurring in the United States each year, a number that is projected to rise as the population ages. In fact, one quarter of adults over the age of 50 will suffer at least one VCF in their lifetime. VCFs cause short term and occasionally long-term pain and disability, and although not immediately life threatening, they are associated with long term mortality. Before the advent of PV, the treatment for VCFs was limited to medical therapy- addressing the pain associated with the fracture but not the fracture itself thus making VCFs practically the only skeletal fracture not treated with orthopedic surgery. Since the introduction of vertebroplasty, over 800 papers, technical notes, and reviews that address this technique have been published with the overwhelming majority reporting significant pain relief and advocating the adoption of the procedure into common practice. Unfortunately, most of these studies had low evidence level and poor scientific design until randomized clinical trials were published in 2009.

Vertebroplasty for refractory back pain (after a period of conservative management of 1 month) constituted the main indication in the overwhelming majority of studies published so far. Although those studies have largely suggested that it does not offer significant improvement in pain or functional status relative to medical therapy or infusion of local anesthesia after this acute phase, the data remains inconclusive and of poor scientific quality. The present study proposes a different rationale: the benefits of vertebroplasty may be occurring in the acute phase (before 1 month) by providing immediate pain relief to the patient, hence allowing early mobilization and preventing medical complications associated with bed rest. In other terms, vertebroplasty may be a first line, acute phase treatment. If the investigators hypothesis holds true, an adequately powered clinical trial may provide sufficient evidence to change the medical indications for vertebroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Presence of:
* at least one and at most two acute VCF (< 6 weeks) at levels caudate to T4, confirmed with physical examination and radiographic imaging
* if timing of the fracture is unclear, the following criteria are required for inclusion in the trial

  1. an MRI scan showing edema at the fracture level(s) or
  2. a bone scan showing increased uptake
* Physical examination showing axial back pain likely secondary to the VCF with restricted mobilization (score not maximum on any one of the following Barthel's Index items: transfer, mobility, bathing, dressing, stairs and toilet use)
* French or English speaking patient willing to return for follow-up or capable of following up with phone interviews if needed

Exclusion Criteria:

* Recent (<30 days) major surgery causing debilitating pain
* Coagulopathy or thrombocytopenia precluding interventional treatment
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Achieving a score of 75 or higher on the Barthel Index functional evaluation score | 30 days after treatment

SECONDARY OUTCOMES:
Rate of cross-over to the alternative treatment | 15 days after treatment
Level of pain as measured by the visual analogue pain scale | at 15 days and 30 days
Proportion of patients located at home | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean Raymond, MD, Principal Investigator — CHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Background] Bourgoin P, Weill A, Tampieri D. CAR Standard for Performance of the Percutaneous Vertebroplasty. Can Assoc Radiol. 2002;(March).
- [Background] Kallmes DF, Comstock BA, Heagerty PJ, Turner JA, Wilson DJ, Diamond TH, Edwards R, Gray LA, Stout L, Owen S, Hollingworth W, Ghdoke B, Annesley-Williams DJ, Ralston SH, Jarvik JG. A randomized trial of vertebroplasty for osteoporotic spinal fractures. N Engl J Med. 2009 Aug 6;361(6):569-79. doi: 10.1056/NEJMoa0900563. PMID 19657122
- [Background] Buchbinder R, Osborne RH, Ebeling PR, Wark JD, Mitchell P, Wriedt C, Graves S, Staples MP, Murphy B. A randomized trial of vertebroplasty for painful osteoporotic vertebral fractures. N Engl J Med. 2009 Aug 6;361(6):557-68. doi: 10.1056/NEJMoa0900429. PMID 19657121
- [Background] Comstock BA, Sitlani CM, Jarvik JG, Heagerty PJ, Turner JA, Kallmes DF. Investigational vertebroplasty safety and efficacy trial (INVEST): patient-reported outcomes through 1 year. Radiology. 2013 Oct;269(1):224-31. doi: 10.1148/radiol.13120821. Epub 2013 May 21. PMID 23696683
- [Background] Voormolen MH, Mali WP, Lohle PN, Fransen H, Lampmann LE, van der Graaf Y, Juttmann JR, Jansssens X, Verhaar HJ. Percutaneous vertebroplasty compared with optimal pain medication treatment: short-term clinical outcome of patients with subacute or chronic painful osteoporotic vertebral compression fractures. The VERTOS study. AJNR Am J Neuroradiol. 2007 Mar;28(3):555-60. PMID 17353335
- [Background] Do HM, Kim BS, Marcellus ML, Curtis L, Marks MP. Prospective analysis of clinical outcomes after percutaneous vertebroplasty for painful osteoporotic vertebral body fractures. AJNR Am J Neuroradiol. 2005 Aug;26(7):1623-8. PMID 16091504
- [Background] Deramond H, Darrason R GP. Percutaneous vertebroplasty with acrylic cement in the treatment of aggressive spinal angiomas. Rachis. 1989;1(2):143-53.
- [Background] Jensen ME, Evans AJ, Mathis JM, Kallmes DF, Cloft HJ, Dion JE. Percutaneous polymethylmethacrylate vertebroplasty in the treatment of osteoporotic vertebral body compression fractures: technical aspects. AJNR Am J Neuroradiol. 1997 Nov-Dec;18(10):1897-904. PMID 9403451
- [Background] Deramond H, Depriester C, Galibert P, Le Gars D. Percutaneous vertebroplasty with polymethylmethacrylate. Technique, indications, and results. Radiol Clin North Am. 1998 May;36(3):533-46. doi: 10.1016/s0033-8389(05)70042-7. PMID 9597071
- [Background] Gangi A, Guth S, Imbert JP, Marin H, Dietemann JL. Percutaneous vertebroplasty: indications, technique, and results. Radiographics. 2003 Mar-Apr;23(2):e10. doi: 10.1148/rg.e10. PMID 12889460
- [Background] Gu YF, Li YD, Wu CG, Sun ZK, He CJ. Safety and efficacy of percutaneous vertebroplasty and interventional tumor removal for metastatic spinal tumors and malignant vertebral compression fractures. AJR Am J Roentgenol. 2014 Mar;202(3):W298-305. doi: 10.2214/AJR.12.10497. PMID 24555629
- [Background] Chen G, Luo ZP, Zhang H, Nalajala B, Yang H. Percutaneous kyphoplasty in the treatment of painful osteoblastic metastatic spinal lesions. J Clin Neurosci. 2013 Jul;20(7):948-50. doi: 10.1016/j.jocn.2012.08.010. Epub 2013 May 3. PMID 23647710
- [Background] Pereira LP, Clarencon F, Cormier E, Rose M, Jean B, Le Jean L, Chiras J. Safety and effectiveness of percutaneous sacroplasty: a single-centre experience in 58 consecutive patients with tumours or osteoporotic insufficient fractures treated under fluoroscopic guidance. Eur Radiol. 2013 Oct;23(10):2764-72. doi: 10.1007/s00330-013-2881-3. Epub 2013 May 21. PMID 23689309
- [Background] Weill A, Chiras J, Simon JM, Rose M, Sola-Martinez T, Enkaoua E. Spinal metastases: indications for and results of percutaneous injection of acrylic surgical cement. Radiology. 1996 Apr;199(1):241-7. doi: 10.1148/radiology.199.1.8633152.
- [Background] Chiras J, Depriester C, Weill A, Sola-Martinez MT, Deramond H. [Percutaneous vertebral surgery. Technics and indications]. J Neuroradiol. 1997 Jun;24(1):45-59. French. PMID 9303944
- [Background] Ruiz Santiago F, Santiago Chinchilla A, Guzman Alvarez L, Perez Abela AL, Castellano Garcia Mdel M, Pajares Lopez M. Comparative review of vertebroplasty and kyphoplasty. World J Radiol. 2014 Jun 28;6(6):329-43. doi: 10.4329/wjr.v6.i6.329. PMID 24976934
- [Background] Yimin Y, Zhiwei R, Wei M, Jha R. Current status of percutaneous vertebroplasty and percutaneous kyphoplasty--a review. Med Sci Monit. 2013 Oct 7;19:826-36. doi: 10.12659/MSM.889479. PMID 24097261
- [Background] Liu J, Li X, Tang D, Cui X, Li X, Yao M, Yu P, Qian X, Wang Y, Jiang H. Comparing pain reduction following vertebroplasty and conservative treatment for osteoporotic vertebral compression fractures: a meta-analysis of randomized controlled trials. Pain Physician. 2013 Sep-Oct;16(5):455-64. PMID 24077192
- [Background] Fotiadou A, Wojcik A, Shaju A. Management of low back pain with facet joint injections and nerve root blocks under computed tomography guidance. A prospective study. Skeletal Radiol. 2012 Sep;41(9):1081-5. doi: 10.1007/s00256-011-1353-6. Epub 2012 Jan 10. PMID 22230900
- [Background] Manchikanti L, Malla Y, Wargo BW, Cash KA, Pampati V, Fellows B. Complications of fluoroscopically directed facet joint nerve blocks: a prospective evaluation of 7,500 episodes with 43,000 nerve blocks. Pain Physician. 2012 Mar-Apr;15(2):E143-50. PMID 22430660
- [Background] Melton LJ 3rd. Epidemiology of spinal osteoporosis. Spine (Phila Pa 1976). 1997 Dec 15;22(24 Suppl):2S-11S. doi: 10.1097/00007632-199712151-00002. PMID 9431638
- [Background] Jones G, White C, Nguyen T, Sambrook PN, Kelly PJ, Eisman JA. Prevalent vertebral deformities: relationship to bone mineral density and spinal osteophytosis in elderly men and women. Osteoporos Int. 1996;6(3):233-9. doi: 10.1007/BF01622740. PMID 8783298
- [Background] Bliuc D, Nguyen ND, Milch VE, Nguyen TV, Eisman JA, Center JR. Mortality risk associated with low-trauma osteoporotic fracture and subsequent fracture in men and women. JAMA. 2009 Feb 4;301(5):513-21. doi: 10.1001/jama.2009.50. PMID 19190316
- [Background] Rousing R, Andersen MO, Jespersen SM, Thomsen K, Lauritsen J. Percutaneous vertebroplasty compared to conservative treatment in patients with painful acute or subacute osteoporotic vertebral fractures: three-months follow-up in a clinical randomized study. Spine (Phila Pa 1976). 2009 Jun 1;34(13):1349-54. doi: 10.1097/BRS.0b013e3181a4e628. PMID 19478654
- [Background] Diamond TH, Bryant C, Browne L, Clark WA. Clinical outcomes after acute osteoporotic vertebral fractures: a 2-year non-randomised trial comparing percutaneous vertebroplasty with conservative therapy. Med J Aust. 2006 Feb 6;184(3):113-7. doi: 10.5694/j.1326-5377.2006.tb00148.x. PMID 16460295
- [Background] Alvarez L, Alcaraz M, Perez-Higueras A, Granizo JJ, de Miguel I, Rossi RE, Quinones D. Percutaneous vertebroplasty: functional improvement in patients with osteoporotic compression fractures. Spine (Phila Pa 1976). 2006 May 1;31(10):1113-8. doi: 10.1097/01.brs.0000216487.97965.38. PMID 16648745
- [Background] Whitley E, Ball J. Statistics review 4: sample size calculations. Crit Care. 2002 Aug;6(4):335-41. doi: 10.1186/cc1521. Epub 2002 May 10. PMID 12225610